CLINICAL TRIAL: NCT06367361
Title: Non-inferiority, Controlled, Randomized, Single-blind Study for Compare Regimens of One and Two Doses of Oxfendazole Versus a Schedule of Two Doses of Triclabendazole to Treat Chronic Fascioliasis
Brief Title: One and Two Doses of Oxfendazole Versus a Schedule of Two Doses of Triclabendazole in Chronic Fascioliasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Oxfendazole Development Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIDISI 201221; U01AI155323 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-04-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Fascioliasis
MeSH Terms: conditions — Fascioliasis | interventions — oxfendazole; Triclabendazole

STUDY DESIGN:
Intervention Model Description: Study arm 1: Oxfendazole 100 mg capsules at 20 mg/kg of body weight as a single oral dose administered with a lipid containing meal under direct observation.
  Study arm 2: Oxfendazole 100 mg capsules at 20 mg/kg of body weight per dose in two oral doses separated 24 hours each administered with a lipid containing meal under direct observation.
  Study arm 3: Triclabendazole 250 mg tablets at 10 mg/kg of body weight per dose in two oral doses separated 24 hours each administered with a lipid containing meal under direct observation.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The laboratory personnel processing the stool microscopy tests will be blinded to the treatment assignment. Thus, the intervention will be blinded to the assessors of the primary endpoint.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oxfendazole single dose (Experimental): Oxfendazole 100 mg capsules at 20 mg/kg of body weight as a single oral dose administered with a lipid containing meal under direct observation.
  Interventions: Drug: Oxfendazole
- Oxfendazole two doses (Experimental): Oxfendazole 100 mg capsules at 20 mg/kg of body weight per dose in two oral doses separated 24 hours each administered with a lipid containing meal under direct observation.
  Interventions: Drug: Oxfendazole
- Triclabendazole (Active Comparator): Triclabendazole 250 mg tablets at 10 mg/kg of body weight per dose in two oral doses separated 24 hours each administered with a lipid containing meal under direct observation.
  Interventions: Drug: Triclabendazole

INTERVENTIONS:
Drug: Oxfendazole — Human studies have shown that doses up to 60 mg/kg (approximately 3.6 g for a 60-kg human, which is considered the average weight of an adult in developing countries) are safe and that repeated doses of 15 mg/kg (approximately 900 mg for a 60-kg human) daily for 5 days are safe. A single dose of OXF results in significant plasma drug concentrations that reach a Cmax plateau after doses of 15 mg/kg.75 The dose to be studied in this trial is 20 mg/kg (1200 mg maximum dose), a dose only slightly higher than that achieving a Cmax plateau. This dose was conservatively selected to account for interindividual variation in plasma levels and deemed well tolerated and safe based on laboratory and ECG evaluations.
  Other Names: Fenbendazole sulfoxide; Synanthic
  Arms: Oxfendazole single dose; Oxfendazole two doses
Drug: Triclabendazole — The standard of care for the treatment of fascioliasis according to the same guidelines is two 10 mg/kg doses of TCBZ 24 hours apart administered with a fat containing meal. The subjects in one of the arms of the study will receive this treatment as the standard of care. Subjects from any of the arms that fail to achieve parasitological cure will receive rescue treatment off the study with two doses of TCBZ as recommended by the Peruvian guidelines.
  Arms: Triclabendazole

SUMMARY:
Randomized clinical trial comparing the efficacy and safety of oxfendazole at 20 mg/kg per dose in one and two dose regimens with a two-dose regimen of triclabendazole at 10 mg/kg in an endemic region of the highlands of Peru. Adults with fascioliasis in rural communities will be screened for inclusion and exclusion criteria and a total of 336 subjects (112 per study arm) with chronic Fasciola infection will be enrolled and assigned randomly to the study arms in a 1:1:1 ratio. The primary efficacy (cure and egg reduction) endpoints will be assessed on day 7 and 30 post treatment. The secondary safety endpoint visits will be performed in days 0, 3, 7 and 30 post-treatment and Population Pharmacokinetics (PK) modeling studies will be performed in the first 24 hours after the first dose of oxfendazole.

DETAILED DESCRIPTION:
Quality Control and Quality Assurance Following a written Data Safety and Monitoring Board (DSMB)-accepted site quality management plan, the participating site and the subcontractors will be responsible for conducting routine quality assurance and quality control activities to internally monitor study progress and protocol compliance. The site principal investigator will provide direct access to all study-related sites, source data/data collection forms, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

The site principal investigator will ensure all study personnel are appropriately trained and applicable documentations are maintained on site. The study principal investigator is the person primarily responsible for assuring compliance. The study principal investigator will regularly review the study progress with team members and conduct periodic audits to ensure that informed consent has been obtained and documented. The principal investigator will review the team operations and progress to ensure that study records are up to date, complete, and kept in a secure place accessible only to appropriate study personnel.

Data Handling and Record Keeping The investigator is responsible to ensure the accuracy, completeness, legibility, and timeliness of the data reported. All source documents will be completed in a neat, legible manner to ensure accurate interpretation of data.

Data collection forms will be derived from the Case Report Forms (CRF) and provided to the study site to record and maintain the data for each subject enrolled in the study. Data reported in the CRF derived from source documents will be consistent with the source documents or the discrepancies will be explained.

The data collection is the responsibility of the clinical trial staff at the site under the supervision of the site principal investigator. The investigator will maintain complete and accurate documentation for the trial. All source documents and laboratory reports will be reviewed by the clinical team and data entry staff to ensure the accuracy and completeness. Adverse Events (AE) will be graded, assessed for severity and causality, and reviewed by the site principal investigator or a designee.

Data Capture Methods Clinical data, including AE and Concomitant Medication (ConMed) and clinical laboratory data will be entered into a pre-designed Electronic Case Report Forms (eCRF) on REDCap. The clinical data will be entered directly from the source documents. The CRF can be considered as a source document.

The access to the REDCap platform will be strictly limited to study staff. The level of access and capabilities for creating new records and changing existing records will be assigned according to specific staff work and need. For example, laboratory staff will only have access to the CRF for reporting test results and not to the CRF where the intervention arm or assigned drug is documented. Laboratory staff will not be able to make changes to any forms except the results form. REDCap's log-in trail will allow the principal investigator to track access to the platform and the changes made to the record during the time logged-in. The platform will be strictly password protected and limited to designated trial personnel. Subjects will be assigned a unique identifier. All subject's records or data sets transferred to the sponsor will contain the identifier only. Subject's names or information that would identify the subject will not be transferred. Quality control will be performed as outlined in Chapter 13 of the protocol. The quality control procedures will be specified in the Manual of Procedures (MoP) and CRF guidance.

Types of Data The data for this trial will include clinical, demographic, safety, hematology and chemistry laboratory values, neuroimaging (MRI) and results of stool egg counts.

Timing/Reports Safety data will be reviewed by the DSMB per the DSMB charter for this trial. The DSMB will review available safety data. Interim statistical reports may be generated as deemed necessary and appropriate by the Division of Microbiology and Infectious Diseases (DMID).

Subjects found to have intestinal parasites in the final stool examination will be contacted and referred to a local health provider to receive standard of care therapy at no cost.

Study Records Retention Study records and reports including, but not limited to, CRF, source documents, Informed Consent Forms (ICF), laboratory test results, and study drug disposition records will be retained for at least 2 years after a marketing application is approved for the study product to treat fascioliasis. If no application is filed or if the application is not approved for the study product, records will be retained until 2 years after the investigation is discontinued and the FDA has been notified. The documents will be retained for a longer period if required by local regulations. ICF for future use will be maintained as long as the sample/specimen exists.

No records will be destroyed without the written consent of the sponsor. It is the responsibility of the sponsor to inform the site principal investigator when these documents no longer need to be retained.

Sample Size Considerations The primary outcome for the study will be the parasitological cure rate of chronic fascioliasis assessed by the qualitative (yes/no) results of the Kato Katz and a Rapid Sedimentation stool tests on Visit Day 30. A subject will be considered cured if the result is negative (0 eggs/gr of stool) at 30 days after treatment. Thus, a binomial response (BR) will be obtained where: If stool microscopy = 0 on Day 30, then BR = 1; otherwise, BR = 0.

The primary analysis will consist of the statistical comparisons between binomial proportions for the single dose Oxfendazole (OXF) arm versus the Triclabendazole (TCBZ) arm and the two dose OXF arm versus the TCBZ arm using the Chi square test statistic with an alpha = 5%. Assuming a cure rate of at least 90% for the single OXF dose arm and at least 90% in the TCBZ arm a sample size of n= 112 per group will be able to exclude an effectiveness difference of > 10% in favor of the TCBZ treatment with 80% power and a difference at five percent level of significance. Similarly, assuming the same effectiveness (at least 90%) for the double OXF dose arm and the TCBZ arm, a sample size of n= 112 per group will be able to exclude an effectiveness difference of > 10% in favor of the TCBZ treatment with 85% power and a difference at five percent level of significance.

Final Analysis Plan The efficacy analysis will be performed in a modified Intention-To-Treat approach. All subjects who were randomized in the study and receive at least one dose of study medication will be considered evaluable and entered in the final analysis database. Subjects in this population will be analyzed according to the group to which they were originally randomized. The same criteria to define the population will be used for the safety analysis. Subjects who do not complete outcome assessments will be considered treatment failures regardless of their randomization group and final status.

Initially, the distribution of baseline population characteristics collected in visit day 1 will be summarized according to the randomization arms using frequencies, means (±SD), medians (interquartile range), and ranges. The characteristics of the groups will be compared using Chi square tests for categorical variables and the T-test (ANOVA if indicated) for the continuous variables. The primary efficacy endpoint will be summarized as the percent of subjects with parasitological cure in each arm at visit day 30. The efficacy between groups will be compared using a Chi Square test with a p ≤ 0.05 to determine the significance off the differences. The efficacy analyses will also be performed using generalized linear regression models to assess any possibility of effect modification and to adjust for any population (study strata/province) and parasitological characteristic that may appeared to be unbalanced after randomization. The egg reduction end point will be analyzed calculating the mean (or median if indicated) egg reduction for the treatment groups and comparing them using the T-Test (or Mann-Whitney test if indicated). Similarly, the egg reduction tests results will be modeled using multiple generalized linear regression to account for imbalances between the groups. Finally, the absolute frequency of all AEs and specifically Serious Adverse Events (SAE) will be compared post-treatment versus baseline using Poisson models for count data to determine potential safety concerns. The proportion of individuals with SAE will be also calculated and compared between arms. A detailed Analysis Plan will be submitted to the Study DSMB for approval before any study activities are initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects eighteen years or older with positive stool microscopy and/or egg counts.
2. Subjects capable of understanding the informed consent process and providing written informed consent.
3. Willingness to give informed consent.

Exclusion Criteria:

1. Subjects reporting previous treatment for fascioliasis
2. Subjects with a stool egg count > 300 eggs/g stool
3. Women with a positive urine pregnancy test or planning to become pregnant
4. Women that are nursing
5. Alanine aminotransferase (ALT) ≥ 3 or Aspartate aminotransferase (AST) ≥ 3 times above the upper limit of normal
6. Subjects with active cerebral cysticercosis determined by serology and imaging studies
7. Subjects with known liver disease, liver cirrhosis, or end stage renal disease
8. Subjects with known allergy or AEs to benzimidazole drugs
9. Subjects taking carbamazepine, phenobarbital, phenytoin, or other medication known to decrease the serum concentrations of benzimidazoles.
10. Women unable or unwilling to use an acceptable birth control method

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Parasitological cure rate of chronic fascioliasis | At day 30 post-treatment.
  The cure rate will be expressed as the proportion of subjects in each arm with negative tests for Fasciola eggs.
Egg reduction rate day 7 | At day 7 post-treatment.
  The egg reduction rate will be expressed as a percentage calculated comparing the visit egg count to the baseline egg count
Egg reduction rate day 30 | At day 30 post-treatment.
  The egg reduction rate will be expressed as a percentage calculated comparing the visit egg count to the baseline egg count

SECONDARY OUTCOMES:
Safety information on day 0 | Day 0 after first dose of study medication.
  Safety information will be collected using a symptoms questionnaire and expressed as the proportion of subjects with adverse events in each arm.
Safety information on day 3 | Day 3 after first dose of study medication.
  Safety information will be collected using a symptoms questionnaire and expressed as the proportion of subjects with adverse events in each arm.
Safety information on day 7 | Day 7 after first dose of study medication.
  Safety information will be collected using a symptoms questionnaire and expressed as the proportion of subjects with adverse events in each arm.
Safety information on day 30 | Day 30 after first dose of study medication.
  Safety information will be collected using a symptoms questionnaire and expressed as the proportion of subjects with adverse events in each arm.
Laboratory safety information day 7 | Day 7 after first dose of study medication
  Safety information will be assessed using laboratory testing and expressed as the proportion of subjects in each arm with abnormal values.
Laboratory safety information day 30 | Day 30 after first dose of study medication
  Safety information will be assessed using laboratory testing and expressed as the proportion of subjects in each arm with abnormal values.
Population pharmacokinetics model constructs for oxfendazole | Day 0
  The plasma levels of oxfendazole will be expressed as a scale using a unit of mass over a unit of volume (micrograms/microliter) and modeled with a population-based approach to assess the disposition and exposure to these drugs forms.
Population pharmacokinetics model constructs for oxfendazole sulfone | Day 0
  The plasma levels of oxfendazole sulfone will be expressed as a scale using a unit of mass over a unit of volume (micrograms/microliter) and modeled with a population-based approach to assess the disposition and exposure to these drugs forms.
Population pharmacokinetics model constructs fenbendazole | Day 0
  The plasma levels of fenbendazole will be expressed as a scale using a unit of mass over a unit of volume (micrograms/microliter) and modeled with a population-based approach to assess the disposition and exposure to these drugs forms.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel M Cabada, MD MSc, Study Chair — University of Texas; Lourdes Rodriguez, MD, Principal Investigator — Asociacion CerviCusco; Hector H Garcia, MD PhD, Study Chair — Universidad Peruana Cayetano Heredia

IPD SHARING:
Plan to Share IPD: No